CLINICAL TRIAL: NCT07297823
Title: Sex Differences in Cold-Induced Changes in Maximal Fat Oxidation: A Pilot Study
Brief Title: Sex Differences in Cold-Induced Changes in Maximal Fat Oxidation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 7231
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Exercise
Keywords: exercise; fat; temperature; cold; metabolism
MeSH Terms: conditions — Motor Activity; Platelet Glycoprotein IV Deficiency; Common Cold | interventions — Cold Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise at room temperature (Active Comparator): Study participants will ride an exercise bike
  Interventions: Other: Room Temperature
- Exercise at cold temperature (Experimental): Study participants will ride an exercise bike. Room temperature will be 5 ºC
  Interventions: Other: Cold temperature

INTERVENTIONS:
Other: Cold temperature — Room temperature will be decreased to 5 ºC
  Arms: Exercise at cold temperature
Other: Room Temperature — Exercise condition for control arm
  Arms: Exercise at room temperature

SUMMARY:
The purpose of this research study is to determine if the cold-induced change in fat burning during exercise is different between females and males.

DETAILED DESCRIPTION:
It is well characterized that females rely more on fat oxidation compared to men during standardized exercise. Exposure to cold during exercise increases fat oxidation in humans. It has been shown that the biological sex differences in substrate oxidation observed during exercise persist in the cold. However, it is unclear if the degree of the effect of cold on substrate oxidation during exercise is different between females and males.

The purpose of this study is to determine if the change in maximal fat oxidation that occurs in cold compared to room temperature environments is different between females and males.

The hypotheses are 1) females will have greater maximal fat oxidation than males in both conditions, and 2) the change in maximal fat oxidation between the control and cold conditions will be the same in females and males.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years (inclusive)
* Weight stable (no change in body mass greater than 5 lbs. within the previous 6 months.
* Willing to abstain from caffeine and alcohol for 24-hours prior to two different study visits
* Competency in English as informally assessed by comprehension of the Informed Consent. This study involves maximal exercise testing; for safety reasons, the ability for clear and rapid communication will be necessary between the research participants and the investigators.
* Regular exercise (i.e., at least 150 minutes of moderate-vigorous exercise per week)

Exclusion Criteria:

* Use of hormonal contraceptives
* History of autonomic, cardio-pulmonary, and/or metabolic disease (including heart failure, hypertension, arrhythmia, vascular disease, and/or diabetes)
* Pregnancy or breast feeding
* Habitual use of tobacco/nicotine products or recreational drugs (2 or more uses within the previous month)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Fat Oxidation | During exercise while in the lab
  Using indirect calorimetry, fat oxidation will be determined. The maximal value for fat oxidation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, Principal Investigator — Colorado State University

IPD SHARING:
Plan to Share IPD: Undecided